CLINICAL TRIAL: NCT01798901
Title: Phase I Study of AR-42 and Decitabine in Acute Myeloid Leukemia
Brief Title: AR-42 and Decitabine in Treating Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alison Walker (Other)
Responsible Party: Sponsor-Investigator, Alison Walker, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-11130; NCI-2013-00122 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-02-22; First posted 2013-02-26 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Recurrent Adult Acute Myeloid Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; AML; AR-42; Decitabine
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myeloid, Acute | interventions — HDAC-42; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (HDAC inhibitor AR-42, decitabine) (Experimental): INDUCTION THERAPY: Patients receive HDAC inhibitor AR-42 PO daily on days 1, 3, and 5 or 1, 3, 4, 5 and decitabine IV over 1 hour on days 6-15. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients achieving CR or CRi receive HDAC inhibitor AR-42 as in Induction Therapy and decitabine IV over 1 hour on days 6-10. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: HDAC inhibitor AR-42; Drug: decitabine; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: HDAC inhibitor AR-42 — Given PO
  Other Names: AR-42
Drug: decitabine — Given IV
  Other Names: 5-aza-dCyd; 5AZA; DAC
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial studies the side effects and best dose of AR-42 when given together with decitabine in treating patients with acute myeloid leukemia. AR-42 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving AR-42 together with decitabine may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the biologic effective and tolerable dose (BETD) of AR-42 (histone deacetylase [HDAC] inhibitor AR-42) in combination with a 10 day schedule of decitabine in acute myeloid leukemia (AML) in adults (Stratum 1) and children (Stratum 2).

II. To define the specific toxicities and the dose limiting toxicity (DLT) of AR-42 in combination with a 10 day schedule of decitabine in adults and children.

SECONDARY OBJECTIVES:

I. To describe biologic activity of the combination of AR-42 and decitabine (changes in micro ribonucleic acid [RNA] [miR]-29b expression; specificity protein 1 [Sp1], deoxyribonucleic acid [DNA] (cytosine-5-)-methyltransferase [DNMT]1, 3A and 3B, KIT and FMS-like tyrosine kinase 3 [FLT3] RNA and protein levels).

II. To provide preliminary data for clinical response with the combination of AR-42 and decitabine in adults and in children.

III. To provide preliminary data on correlation of biologic endpoints and clinical response (particularly miR-29b expression).

OUTLINE: This is a dose-escalation study of HDAC inhibitor AR-42.

INDUCTION THERAPY: Patients receive HDAC inhibitor AR-42 orally (PO) daily on days 1, 3, and 5 or 1, 3, 4, 5 and decitabine intravenously (IV) over 1 hour on days 6-15. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients achieving complete remission (CR) or morphologic CR with incomplete blood count recovery (CRi) receive HDAC inhibitor AR-42 as in Induction Therapy and decitabine IV over 1 hour on days 6-10. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (stratum 1) must be age >= 18 with relapsed or refractory acute myeloid leukemia (AML) or age >= 60 with previously untreated AML who are not candidates for or refuse standard/conventional induction chemotherapy (e.g. the 7+3 combination of cytarabine and an anthracycline); pediatric patients, age 3 to < 18 years (stratum 2) will be eligible with AML in second relapse or with refractory disease
* Patients with secondary AML or therapy related disease (t-AML) are eligible
* Patients who received decitabine or 5-azacitidine as prior treatment for myelodysplastic syndrome (MDS) (or AML) remain eligible for the dose escalation phase of the study; however, neither of these agents is permitted within 3 months of study entry; patients who have received prior decitabine or 5- azacitidine will be excluded from the expansion phase of the trial
* If the patient has co-morbid medical illness, life expectancy attributed to this must be greater than 6 months
* Performance status: Adults (>= 18 years) must be Eastern Cooperative Oncology Group (ECOG) performance status =< 2; pediatric patients (< 18 years) must be at least Lansky > 50%
* Total bilirubin < 2.0 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 X institutional upper limit of normal
* Creatinine < 2.0 mg/dL (adults > 18 years); < 1.3 x upper limit normal for age (pediatric patients < 18 years)
* New York Heart Association (NYHA) congestive heart failure (CHF) class II or better
* The effects of decitabine and AR-42 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason, both men and women must agree to use adequate contraception (barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; if the patient does not agree, the patient is not eligible; should a woman become pregnant or suspect she is pregnant while participating in the study, she should inform her treating physician immediately
* Ability to understand and willingness to sign the written informed consent document
* Patients must have recovered from the toxicity of prior therapy to less than grade 2

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study; hydroxyurea may be administered for control of leukocytosis both pre-treatment and during cycle 1 only
* Patients receiving any other investigational agents or patients that have received other investigational agents within 28 days of enrollment
* Patients with active central nervous system disease or with a single granulocytic sarcoma as sole site of disease
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to decitabine or AR-42 that cannot be managed with oral antihistamines, antipyretics (ie. acetaminophen) or low dose corticosteroids (< 10 mg oral prednisone or equivalent corticosteroid)
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; as infection is a common feature of AML, patients with active infection are permitted to enroll provided that the infection is under control; myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, uncontrolled hypertension, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Patients with serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Patients with a known confirmed diagnosis of human immunodeficiency virus (HIV) infection (due to concern for increased toxicity with the regimen in combination with highly active antiretroviral therapy [HAART])
* Patients with a known diagnosis of chronic hepatitis B infection (ie. persistence of hepatitis B surface antigen in the blood for 6 months or longer) or a diagnosis of hepatitis C (ie. the presence of anti-hepatitis C (hepatitis C virus [HCV]) antibodies in the peripheral blood) are excluded; patients with a recent diagnosis (< 6 months) of active viral hepatitis B or C are excluded
* Patients who have advanced malignant solid tumors at the time of consideration for enrollment on this trial are excluded; patients who have a history of an advanced malignant solid tumor, but have no evidence of disease at the time of consideration for enrollment, are eligible
* Patients with a known impairment of gastrointestinal (GI) function due to a GI disease such as inflammatory bowel disease (Crohn's disease, ulcerative colitis) or celiac disease, that may significantly alter the absorption of AR-42 are excluded
* Pregnant women or women who are breastfeeding are excluded from this study; confirmation that the subject is not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening; pregnancy testing is not required for post-menopausal or surgically sterilized women
* Diagnosis of prolonged QT syndrome
* Patients with a mean corrected QT interval (QTc) > 450 msec in males and > 470 msec in females
* Inability to swallow capsules

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-09-17 (Actual); Primary Completion 2015-02-19 (Actual); Study Completion 2015-02-19 (Actual)

PRIMARY OUTCOMES:
BETD (biologic effective and tolerable dose) of HDAC inhibitor AR-42, defined as a doubling in miR-29b levels from baseline | Up to 28 days
Maximum tolerated dose (MTD) based on incidence of dose-limiting toxicity (DLT) graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0 | Up to 28 days
Incidence of adverse events, graded according to the NCI CTCAE v4.0 | Up to 3 years
  Toxicities will be tabulated by dose level and summarized in addition to assessing the incidence of DLTs. Severe (grade 3+) toxicities will be summarized by type as well as in summary format of hematologic vs. non-hematologic severe toxicity incidence. DLT-level toxicities will also be summarized and tracked beyond the first cycle of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Walker, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio

REFERENCES:
- [Derived] Cheng H, Xie Z, Jones WP, Wei XT, Liu Z, Wang D, Kulp SK, Wang J, Coss CC, Chen CS, Marcucci G, Garzon R, Covey JM, Phelps MA, Chan KK. Preclinical Pharmacokinetics Study of R- and S-Enantiomers of the Histone Deacetylase Inhibitor, AR-42 (NSC 731438), in Rodents. AAPS J. 2016 May;18(3):737-45. doi: 10.1208/s12248-016-9876-3. Epub 2016 Mar 4. PMID 26943915
- [Derived] Bernot KM, Siebenaler RF, Whitman SP, Zorko NA, Marcucci GG, Santhanam R, Ahmed EH, Ngangana M, McConnell KK, Nemer JS, Brook DL, Kulp SK, Chen CS, Frankhouser D, Yan P, Bundschuh R, Zhang X, Dorrance AM, Dickerson KE, Jarjoura D, Blum W, Marcucci G, Caligiuri MA. Toward personalized therapy in AML: in vivo benefit of targeting aberrant epigenetics in MLL-PTD-associated AML. Leukemia. 2013 Dec;27(12):2379-82. doi: 10.1038/leu.2013.147. Epub 2013 May 10. No abstract available. PMID 23660685
- See also: The Jamesline — http://cancer.osu.edu